CLINICAL TRIAL: NCT02533245
Title: Effect of an Exercise Training Intervention on Health-related Quality of Life and Psychosocial and Behavioral Variables in Adult Solid Organ Transplant Recipients: a Quasi-experimental Study Design
Brief Title: Transplantoux Health Evaluation Study
Acronym: THES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: THES1
Record Dates: First submitted 2015-08-19; First posted 2015-08-26 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Quality of Life
Keywords: Exercise Training; Quality of Life; Patient Reported Outcomes; Organ Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tx exercise group (Experimental): Convenience sample of solid organ transplant recipients (heart, kidney, lung, liver, pancreas, small bowel) participating in the Transplantoux exercise training intervention.
  Intervention:
  * Home-based individualized exercise training program
  * Supervised group training sessions
  * Climb of the Mont Ventoux
  Interventions: Other: Home-based indiviualized exercise training program; Other: Supervised group training sessions; Other: Climb of the Mont Ventoux
- Tx matched control group (No Intervention): Controls are retrieved from the Leuven University Hospital heart, kidney, lung, liver, pancreas, small bowel transplant database and matched (1:4 matching) based on type of transplant, gender, age and time since transplant.
- Healthy exercise group (Experimental): Convenience sample of health care providers (e.g. doctor, paramedic or medical companion involved in care programs for organ Tx) and patient's family members and friends participating in the Transplantoux exercise training intervention.
  Intervention:
  * Supervised group training sessions
  * Climb of the mont ventoux
  Interventions: Other: Supervised group training sessions; Other: Climb of the Mont Ventoux

INTERVENTIONS:
Other: Home-based indiviualized exercise training program — Based on these results of the cardiopulmonary exercise test (CPET) on a cycle ergometer, an individualized training program (cycling/hiking) is prescribed by a physical therapist for 6 months (3x/week, ≥30min/session).
  Arms: Tx exercise group
Other: Supervised group training sessions — 7 supervised group training sessions (cycling/hiking) are organized by a physiotherapist
  Arms: Healthy exercise group; Tx exercise group
Other: Climb of the Mont Ventoux — Cycle or hike up the Mont Ventoux (25.7 km, average slope 4.5%)
  Arms: Healthy exercise group; Tx exercise group

SUMMARY:
The primary aim is to evaluate the short- and long-term effect of the 'Transplantoux' exercise training intervention in solid organ transplant recipients with matched control sample of transplant recipients in view of selected Patient Reported Outcomes (PRO), i.e. health-related quality-of-life (HRQOL), psychosocial and behavioral variables, using a quasi-experimental design.

DETAILED DESCRIPTION:
During the last decades advances in solid organ transplantation, like e.g. organ preservation, surgical techniques and immunosuppressive treatment have contributed to improvements in postoperative survival. Thereby, solid organ transplantation (Tx) has moved from experimental treatment towards a clinical reality and a life-saving surgery, offering most patients a good long-term survival. However, further improvement in long-term survival remains a major challenge.

It is increasingly recognized that non-pharmacological interventions hold the potential to improve long-term outcomes in transplantation as evidence shows that health behavior has been independently associated with transplant outcome (e.g. physical activity, non-smoking, medication adherence). Furthermore, exercise training interventions show positive outcome in a number of populations and limited research in transplantation shows positive outcomes in view of exercise capacity, muscle strength, cardiopulmonary variables and body composition. However, there is a lack of research that evaluates exercise training interventions in view of patient reported outcomes (PROs) in transplant recipients.

In the University Hospitals of Leuven (Belgium) a project named 'Transplantoux' has been launched to enhance physical activity and exercise capacity in transplant recipients. Transplant recipients participate in the 'Transplantoux' exercise training intervention for 6-months with the ultimate goal to cycle or hike up the Mont Ventoux (France) (distance: 25.9 km, mean slope: 4.4%). Extending on a previous safety feasibility study in which we demonstrated that selected Transplant recipients can safely participate in an intense exercise program and that exercise capacity was significantly improved after training. The primary aim of the current study is to evaluate the short- and long-term effect of the 'Transplantoux' intervention in view of selected Patient Reported Outcomes (PROs), i.e. perceived health-related quality-of-life, depressive symptomatology, stress and well-being, physical activity, social contacts and social support, and barriers and motivators to exercise.

The Transplantoux Health Evaluation Study (THES) uses a quasi-experimental design with three convenience samples: 1) a convenience sample of solid organ transplant (Tx)-recipients participating in the Transplantoux exercise training intervention, 2) matched control sample of Tx-recipients not participating in the Transplantoux exercise intervention, and 3) and a convenience sample of healthy controls participating in the Transplantoux exercise intervention. Selected PROs will be assessed using validated self-reported questionnaire. Data collection will be performed at baseline, 3 months (in the middle of the training intervention), 6 months (immediately following the intervention), 9 months (3 months follow-up period) and 12 months (6 months follow-up period).

ELIGIBILITY:
1. Tx exercise group:

   Inclusion Criteria:
   * Tx recipient (heart, lung, liver, kidney, pancreas or small bowel)
   * Age between 18 - 70 years
   * More than 1y post-transplant

   Exclusion Criteria:
   * Rejection last 6 months
   * Severe co-morbidity
   * Contra-indication for severe exercise (e.g. cardiovascular disease)
   * Insufficient knowledge of Dutch language
2. Tx matched control group

   Inclusion Criteria:
   * Tx recipient (heart, lung, liver, kidney, pancreas or small bowel)
   * Age between 18 - 70 years
   * More than 1y post-transplant

   Exclusion Criteria:
   * Rejection last 6 months
   * Insufficient knowledge of Dutch language
3. Healthy exercise group:

Inclusion Criteria:

* Age between 18 - 70 years

Exclusion Criteria:

* Contra-indication for severe exercise
* Insufficient knowledge of Dutch language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in PROs (i.e. perceived quality of life, depressive symptomatology, stress and well-being, physical activity, and social contacts and support) in the Tx exercise group compared with Tx matched control group | baseline, 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Change in PROs (i.e. perceived quality of life, depressive symptomatology, stress and well-being, physical activity, and social contacts and support) in Tx exercise group compared with healthy exercise group | baseline, 3, 6, 9 and 12 months
Compare PROs (i.e. perceived quality of life, depressive symptomatology, stress and well-being, physical activity, and social contacts and support) of the three groups with a representative sample of the Belgian population | baseline
Compare perceived barriers and motivators for physical exercise/activity in the three groups | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Diethard Monbaliu, MD, PhD, Principal Investigator — University Hospital Leuven, Abdominal Transplant Surgery
Locations (1):
- University Hospitals Leuven, Leuven, Belgium